CLINICAL TRIAL: NCT03703323
Title: Comparison of Mortality Impact of Coagulation Rotative Thromboelastometry Analysis Versus Standard Analysis (Prothrombin Ratio) for Patients With Digestive Hemorrage
Brief Title: Comparison of Mortality Impact of Coagulation Rotative Thromboelastometry Analysis Versus Standard Analysis
Acronym: HD-ROTEM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: pandemic situation
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-03-CHRMT
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-01

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rotative thromboelastometry analysis (Experimental): Evaluation of diagnostic properties of coagulation by rotative thromboelastometry in patient with digestive hemorrhage in predictive value of mortality.
  Interventions: Other: Rotative thromboelastometry analysis

INTERVENTIONS:
Other: Rotative thromboelastometry analysis — Obtaining blood sample (one tube of blood)

SUMMARY:
Digestive hemorrhage is a common cause of acute hemorrhage in France, and its mortality remains high despite improvement of endoscopy technique and therapeutics. Hemostasis disorders are an important issue in the patient care both in severity diagnostic and therapeutic plan.

DETAILED DESCRIPTION:
Standard technique of coagulation analysis (prothrombin ratio, activated partial thromboplastin time, fibrinogen and platelet count) do not provide to guide practitioner in reanimation of hemostatic patients in particular when coagulation defect preexisting to the digestive hemorrhage.

In this respect, the main objective of this study is to evaluate the interest of rotative thromboelastometry in the care of patient with digestive hemorrhage and its mortality impact.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patient in reanimation unit or continuous monitoring for digestive hemorrhage before or immediately after digestive endoscopy
* Digestive hemorrhage diagnostic: melena and/or rectal bleeding and/or hematemesis
* Affiliation to the social security
* Have signed an informed consent

Exclusion Criteria:

* Pregnant or nursing woman
* Without digestive fibroscopy
* With an anticoagulant treatment
* With a congenital coagulopathy
* Decision of therapeutic limitation or moribund patient
* With a digestive hemorrhage after an hospitalisation in reanimation unit for an other reason
* Participation in an other study in previous 30 days
* Under trusteeship, guardianship or judicial safeguards

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Mortality | day 28
  28-day mortality rate

SECONDARY OUTCOMES:
Fresh-frozen plasma | day 2
  Number of fresh-frozen plasma used within the first 48 hours of the care
Length of stay | day 28
  Lenght of stay in reanimation unit
Recurrent bleeding | Day 2
  recurrent bleeding within the first 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, France